CLINICAL TRIAL: NCT04832100
Title: A Clinical Approach to Validate the Biological Significance of LPC16:0 as a Discriminating and Pathogenic Biomarker of Fibromyalgia
Brief Title: Bio-significance of LPC16:0 in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-G(I)-20170012
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia, Primary; Pain; Soreness, Muscle; Oxidative Stress; Metabolomics; Lipidomics
Keywords: lysophosphotidylcholine; fibromyalgia; pain; soreness; metabolomics
MeSH Terms: conditions — Fibromyalgia; Pain; Myalgia | interventions — Pregabalin; Imipramine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collection of blood samples for metabolomic and genetic investigations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary fibromyalgia: Adults with complaints of chronic widespread pain at the outpatient department of KMUH were consecutively enrolled over a 5-year period from June 2021 to June 2026. Participants were interviewed by experienced neurologists , and those who fulfilled the 2011 American College of Rheumatology (ACR) criteria for FM were recruited .
  Interventions: Drug: Pregabalin 150mg, imipramine 25mg
- Healthy controls: Age- and sex-matched subjects without pain and soreness were also prospectively recruited as healthy controls.

INTERVENTIONS:
Drug: Pregabalin 150mg, imipramine 25mg — Conventional treatment for fibromyalgia was given to patients. Clinical follow-ups with questionnaires and interview were arranged then.
  Groups: Patients with primary fibromyalgia

SUMMARY:
Fibromyalgia (FM) is a very common but mysterious pain disorder characterized by chronic widespread muscular pain. Fatigue, anxiety and depression are common comorbidities. The syndrome is commonly associated with several symptoms, including fatigue, sleeping disturbance, cognitive impairment, and comorbid pain syndrome, especially irritable bowel symptoms and temporomandibular disease. Anxiety and depression are common psychiatric co-morbidies. Daily stress is believed to trigger or aggravate pain conditions. These symptoms can markedly affect patients' quality of life, and even lead to disability. So far, the etiology and pathogenesis are largely unknown, and diagnostic biomarkers and curative treatment remain to be developed. Recent technological advances enable scientists to explore mechanisms by genetic, transcriptomic, proteomic, and metabolomic researches. However, no definitive result has been concluded for clinical practice so far.

In this study, the investigators use tailored questionnaires to evaluate fibromyalgia and associated symptoms, including numeric rating scale for soreness, widespread soreness index, Fibromyalgia impact questionnaire, Hospital Anxiety and Depression Scale, and perceived stress scale. The investigators also use metabolomics and lipidomic approach to probe the potential pathophysiology of fibromyalgia. In our prior translation research (PMID: 32907805), the investigators found that excessive LPC16:0 resulting from lipid oxidization inflicts psychological stress-induced chronic non-inflammatory pain via activating ASIC3. In this content, our prior translational research identified a potential nociceptive ligand that causes fibromyalgia symptoms, which is likely to function as biomarkers for diagnosis or disease monitor. In the current clinical investigation, the investigators aim to reversely translate the novel findings in animal studies and validate the bio-significance of LPC16:0 for fibromyalgia with clinical approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of fibromyalgia

Exclusion Criteria:

1. Systemic rheumatological or immune disorders (e.g., systemic lupus erythematosus, inflammatory myositis),
2. Systemic use of corticosteroids,
3. Pregnancy,
4. Chronic diseases under poor control
5. Malignancies.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient group: participants with primary fibromyalgia Control group: healthy controls
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire: Numeric rating scale (NRS) for pain and soreness | Changes from baseline NRS at 2 weeks are assessed
  assessment of pain and soreness severity. Score: 0(no symptom) ~10 (worst symptom)
Questionnaire: Numeric rating scale (NRS) for pain and soreness | Changes from baseline NRS at 4 weeks are assessed
  assessment of pain and soreness severity. Score: 0(no symptom) ~10 (worst symptom)
Questionnaire: widespread pain index and widespread soreness index | Change from baseline widespread index at 2 weeks are assessed
  assessment of pain and soreness diffuseness. Score: 0(no symptom) ~19 (mostly diffused symptom)
Questionnaire: widespread pain index and widespread soreness index | Change from baseline widespread index at 4 weeks are assessed
  assessment of pain and soreness diffuseness. Score: 0(no symptom) ~19 (mostly diffused symptom)
Questionnaire: Fibromyalgia impact questionnaire (FIQR) | Change from baseline FIQR at 2 weeks are assessed
  assessment of fibromyalgia impacts and disease severity. Score: 0(no symptom) ~100 (worst symptom)
Questionnaire: Fibromyalgia impact questionnaire (FIQR) | Change from baseline FIQR at 4 weeks are assessed
  assessment of fibromyalgia impacts and disease severity. Score: 0(no symptom) ~100 (worst symptom)
Questionnaire: Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS at 2 weeks are assessed
  assessment of psychological distress. Score: 0 (no symptom) ~42 (worst symptom)
Questionnaire: Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS at 4 weeks are assessed
  assessment of psychological distress. Score: 0 (no symptom) ~42 (worst symptom)
Questionnaire: The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline PSQI at 2 weeks are assessed
  assessment of sleep quality. Score: 0 (no symptom) ~21 (worst sleep quality)
Questionnaire: The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline PSQI at 4 weeks are assessed
  assessment of sleep quality. Score: 0 (no symptom) ~21 (worst sleep quality)
Questionnaire: Perceived stress scale (PSS) | Change from baseline PSS at 2 weeks are assessed
  assessment of perceived stress loading. Score: 0 (no stress) ~40 (highest stressed level)
Questionnaire: Perceived stress scale (PSS) | Change from baseline PSS at 4 weeks are assessed
  assessment of perceived stress loading. Score: 0 (no stress) ~40 (highest stressed level)
Metabolomics investigation | Change from baseline metabolomics at 3 months are assessed
  Laboratory investigation of metabolomic expression, including lactate, creatine, malondialdehyde, protein carbonyls and amino acids.
Lipidomics investigation | Change from baseline metabolomics at 3 months are assessed
  Laboratory investigation of lipidomic expression, including phosphocholine, sphingomyelin, lysophosphatidylcholine and ceramide.
Metabolomics investigation | Change from baseline metabolomics at 6 months are assessed
  Laboratory investigation of metabolomic expression, including lactate, creatine, malondialdehyde, protein carbonyls and amino acids.
Lipidomics investigation | Change from baseline metabolomics at 6 months are assessed
  Laboratory investigation of lipidomic expression, including phosphocholine, sphingomyelin, lysophosphatidylcholine and ceramide.
Metabolomics investigation | Change from baseline metabolomics at 9 months are assessed
  Laboratory investigation of metabolomic expression, including lactate, creatine, malondialdehyde, protein carbonyls and amino acids.
Lipidomics investigation | Change from baseline metabolomics at 9 months are assessed
  Laboratory investigation of lipidomic expression, including phosphocholine, sphingomyelin, lysophosphatidylcholine and ceramide.
Metabolomics investigation | Change from baseline metabolomics at 12 months are assessed
  Laboratory investigation of metabolomic expression, including lactate, creatine, malondialdehyde, protein carbonyls and amino acids.
Lipidomics investigation | Change from baseline metabolomics at 12 months are assessed
  Laboratory investigation of lipidomic expression, including phosphocholine, sphingomyelin, lysophosphatidylcholine and ceramide.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Raw and analyzed data will be shared upon written request to the corresponding author from any qualified investigator.

REFERENCES:
- [Derived] Hung CH, Tsai MH, Wang PS, Liang FW, Hsu CY, Lee KW, Fong YO, Han DS, Lee CH, Lai CL, Chen CC. Oxidative stress involves phenotype modulation of morbid soreness symptoms in fibromyalgia. RMD Open. 2023 Mar;9(1):e002741. doi: 10.1136/rmdopen-2022-002741. PMID 36918228

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04832100/Prot_SAP_000.pdf